CLINICAL TRIAL: NCT05051930
Title: Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Primary Efficacy of TQC3721 Suspension for Inhalation
Brief Title: A Clinical Trial of TQC3721 Suspension for Inhalation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC3721-I-01
Record Dates: First submitted 2021-08-17; First posted 2021-09-21 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQC3721 suspension for inhalation (Experimental): Participants will receive 0.2 mg/1.0 mg/3.0 mg/6.0 mg/12.0 mg/24.0 mg single dose of TQC3721 suspension for inhalation on Day 1.
  Interventions: Drug: TQC3721 suspension for inhalation
- TQC3721 suspension placebo for inhalation (Placebo Comparator): Participants will receive 0mg single dose of TQC3721 suspension placebo for inhalation on Day 1.
  Interventions: Drug: TQC3721 suspension placebo for inhalation

INTERVENTIONS:
Drug: TQC3721 suspension for inhalation — Participants will receive 0.2 mg/1.0 mg/3.0 mg/6.0 mg/12.0 mg/24.0 mg single dose of TQC3721 suspension for inhalation.
  Arms: TQC3721 suspension for inhalation
Drug: TQC3721 suspension placebo for inhalation — Participants will receive 0mg single dose of TQC3721 suspension placebo for inhalation .
  Arms: TQC3721 suspension placebo for inhalation

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetic characteristics of TQC3721 suspension for inhalation in single/multiple administration(s) in healthy subjects; to evaluate the safety,tolerability and efficacy TQC3721 suspension for inhalation in multiple administrations in patients with Chronic Obstructive Pulmonary Disease（COPD）and asthma.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before the trial, fully understand the content, process and possible adverse reactions of the test;
* Able to complete the study according to the requirements of protocol;
* Aged between 18 and 65 years old, both men and women;
* For healthy subjects: Male ≥50kg, female ≥45kg,body mass index(BMI)=weight (kg)/height 2 (m2), BMI is 18-28 kg/m2 (including the critical value); For patients: BMI is 18-28 kg/m2 (including the critical value), and body weight is ≥45kg.
* For healthy subjects: normal or abnormal vital signs, physical examination, laboratory examination, electrocardiogram, and imageological examination have no clinical significance;
* For healthy subjects: FEV1 and forced vital capacity(FVC) are at least 90% of the predicted values;
* Subjects (including male subjects) have no pregnancy plan and have voluntarily taken effective contraceptive measures for at least 1 month after being screened to the last use of the study drug;
* For patients: Vital signs range: systolic blood pressure 90 to 140mmHg, diastolic blood pressure 50 to 90 mmHg, heart rate 50 to 90 bpm;
* For patients: 12-lead electrocardiogram with QT interval corrected ≤450 msec (males) or ≤470 msec (females), QRS interval ≤120 msec, PR interval ≤200 msec and no morphologic and other clinical significant abnormalities (such as left band branch block, atrioventricular node dysfunction, ischemic ST segment abnormalities);
* For patients: Ability to perform acceptable and reproducible spirometry;
* For patients: According to the diagnostic criteria of 2018 Practical Edition of Guidelines for the Diagnosis and Treatment of COPD, the patient was diagnosed with COPD for at least 1 year;Post-bronchodilator spirometry at screening must demonstrate FEV1/FVC ratio of ≤0.70 and FEV1 must be ≥40 % to ≤80% of predicted normal;
* For patients: mMRC Scoring at screening ≥2;
* For patients: Clinically stable COPD in the previous 4 weeks;
* For patients: Capable of withdrawing long acting bronchodilators until the end of the treatment period, and short acting bronchodilators for 8 hours prior to administration of study medication;
* For patients: Current and former smokers with a smoking history of ≥10 pack years（smoking at least 20 cigarettes a day for 10 years or at least 10 cigarettes a day for 20 years）;
* For patients: beta agonists are currently used only "when needed";
* For patients: Never smoked or An ex-smoker for ≥6 months；

Exclusion Criteria:

* Preexisting or existing the neuropsychiatric system, respiratory system, cardiovascular system, digestive system, hemo-lymphatic system, immune system, liver and kidney dysfunction, endocrine system, musculoskeletal system, or other disease that the investigator assesses that may affect drug metabolism or safety.
* For healthy subjects: Have a history of fainting needles, fainting blood.
* For healthy subjects: Known allergy to the study drug and their metabolites or any of the excipients of the formulation.
* For healthy subjects: Those who smoked more than 5 cigarettes per day during the 3 months before the trial.
* A history of alcohol abuse in the past 6 months (14 units of alcohol consumed per week: 1 unit =360 ml of beer or 45 ml of 40% alcohol spirits or 150 ml of wine).
* For healthy subjects: Donated blood or had substantial loss of blood (more than 400 mL) within 2 months before the test.
* For healthy subjects: Had taken any prescription, over-the-counter, vitamin product or herbal medicine within 1 month prior to the use of the study drug.
* Participated in other clinical trials within 3 months prior to this study.
* Positive for hepatitis (including hepatitis B and C), human immunodeficiency virus（HIV） or syphilis at screening.
* Women who are pregnant or breast-feeding.
* Positive test for alcohol.
* For healthy subjects: Blood collection is difficult or cannot tolerate venipuncture blood collection.
* For healthy subjects: The subject is unable or can not comply with ward management regulations.
* For healthy subjects: The subject is unable to complete the study due to personal reasons.
* For healthy subjects: Any circumstances that the investigator considers to pose a safety risk to the subject during the study or may interfere with the conduct of the study.
* For patients: Intolerance to salbutamol, tiotropium, or this product or prior exposure to Ensifentrine (RPL554).
* For patients: Use of any medicine within 4 weeks prior to initiation of the study drug, including non-prescription medications and herbs, except vitamins.
* For patients: Physical examination findings that researchers consider clinically significant at the time of screening.
* For patients: A history of cardiovascular disease (including arrhythmias) or active hyperthyroidism.
* For patients: History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localised basal cell carcinoma of the skin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | From the enrollment of the subjects to 72 hours after the last administration
  The Number of adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Incidence of adverse events | From the enrollment of the subjects to 72 hours after the last administration
  The Incidence of adverse events as assessed by CTCAE v5.0
Number of adverse events related to the study drug | From the enrollment of the subjects to 72 hours after the last administration
  The number of adverse events associated with the study drug assessed by CTCAE V5.0
Incidence of adverse events associated with the study drug | From the enrollment of the subjects to 72 hours after the last administration
  Incidence of adverse events associated with the study drug as assessed by CTCAE V5.0
Area Under The Curve（AUC） | Within 60 minutes before each administration, to 72 hours after administration
  Area under the curve
Plasma drug peak concentration（Cmax ） | Within 60 minutes before each administration, to 72 hours after administration
  Plasma drug peak concentration
Time to peak（Tmax） | Within 60 minutes before each administration, to 72 hours after administration
  Time to maximum concentration following drug administration

SECONDARY OUTCOMES:
Elimination half-life time（t1/2） | Within 60 minutes before each administration, to 72 hours after administration
  Apparent terminal elimination half-life following drug administration
Apparent volume of distribution（Vd） | Within 60 minutes before each administration, to 72 hours after administration
  Apparent volume of distribution
Clearance（CL） | Within 60 minutes before each administration, to 72 hours after administration
  Clearance
Forced Expiratory Volume in the first second (FEV1) for patients with Chronic Obstructive Pulmonary Disease（COPD） or asthma | From before administration to 3 hours after administration
  Mean Change From Baseline in Peak FEV1 (Over 3 Hours)
Mean Change From Baseline FEV1 to Morning Trough FEV1 | From the enrollment of the subjects to to 72 hours after administration
  Mean Change From Baseline FEV1 to Morning Trough FEV1
Mean Change From Baseline FEV1 to Average FEV1 | From the enrollment of the subjects to to 72 hours after administration
  Mean Change From Baseline FEV1 to Average FEV1
COPD Assessment Test (CAT) for patients with COPD | From enrollment to 4 weeks after administration
  Mean Change From Baseline in COPD Assessment Test (CAT) Scoring at Week 4.The score range is 0 to 40 (0 to 10 is minor influence;11 to 20 is moderate; 21 to30 is severe;31 to 40 is very severe), and more than 10 indicates more symptoms.
Modified medical research council(mMRC) for patients with COPD or asthma | From enrollment to 4 weeks after administration
  Mean Change From Baseline in mMRC Scoring at Week 4.The severity is measured on a five-point scale from 0 to 4, with a higher score indicating more severe respiratory distress.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China